CLINICAL TRIAL: NCT06127693
Title: The Roles of Childhood Adversity and Inflammatory Reactivity in Promoting Pain and Fatigue After Provocation
Brief Title: Childhood Adversity, Inflammatory Reactivity and Persistent Pain
Acronym: CAIR
Status: Completed | Type: Observational
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Victoria Madden, Associate Professor, University of Cape Town
Other Study IDs: HREC REF 560/2021
Record Dates: First submitted 2023-10-31; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain; Central Sensitisation; Immune Response; Adverse Childhood Experiences
Keywords: Secondary hyperalgesia; Pain; Innate immune response; Adverse childhood experiences; Conditioned pain modulation
MeSH Terms: conditions — Chronic Pain; Hyperalgesia; Pain | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild childhood adversity (control): Score of 25-36 on the Childhood Trauma Questionnaire-short form.
  Interventions: Drug: Tetravalent Influenza Vaccine; Behavioral: High-frequency electrical stimulation
- Moderate childhood adversity: Score of 37-67 on the Childhood Trauma Questionnaire-short form.
  Interventions: Drug: Tetravalent Influenza Vaccine; Behavioral: High-frequency electrical stimulation
- Severe childhood adversity: Score of >67 on the Childhood Trauma Questionnaire-short form.
  Interventions: Drug: Tetravalent Influenza Vaccine; Behavioral: High-frequency electrical stimulation

INTERVENTIONS:
Drug: Tetravalent Influenza Vaccine — All participants will receive the tetravalent influenza vaccine
  Other Names: flu vaccine
Behavioral: High-frequency electrical stimulation — All participants will receive High-frequency electrical stimulation

SUMMARY:
The goal of this observational study is to investigate how adverse experiences during childhood are linked to people experiencing persistent pain and fatigue in adulthood.

The questions the investigators aim to answer are:

1. Does participant-reported childhood adversity predict levels of IL-6 and TNF-α after in vitro provocation of whole blood using endotoxin?
2. Do levels of IL-6 and TNF-α after in vitro immune provocation using endotoxin predict vulnerability to persistent pain and fatigue after in vivo immune provocation (tetravalent influenza vaccine)?
3. Do levels of IL-6 and TNF-α after in vitro immune provocation using endotoxin predict vulnerability to persistent pain and fatigue after in vivo neural provocation?

For this study, the investigators will recruit and enrol 96 healthy human adults (18 - 65 years old) with a range of adverse experiences during childhood. Participants will attend 2 study sessions during which the investigators will take a sample of blood, assess pressure pain threshold before and after cold water immersion, assess heart rate variability, and assess the surface area of secondary skin hypersensitivity after electrical stimulation. At the end of the first session, participants will receive the influenza vaccination.

DETAILED DESCRIPTION:
Background

Adverse experiences during childhood (childhood adversity) are associated with an increased risk of persistent pain and fatigue in adulthood. While the physiological relationships that link childhood adversity, persistent pain, and fatigue are unclear, all three factors are each associated with heightened innate immune and neural responses in adulthood. As such, neuroimmune interactions could underlie the relationship between childhood adversity, persistent pain, and fatigue, although the balance between the immune and neural influences likely varies across individuals.The investigators hypothesise that childhood adversity influences persistent pain and fatigue by priming: 1) immune, 2) neural, or 3) both systems, within an individual. Although previous studies have examined either immune or neural processes representing vulnerability to persistent pain and fatigue, the investigators are not aware of any study that has investigated both systems in the same cohort.

Methods

96 healthy adult humans with a range of childhood adversity history will undergo psychophysical testing before and after in vivo neural provocation (high frequency electrical stimulation) and, separately, immune provocation (influenza vaccine). Study proxies for vulnerability to persistent pain are surface area of secondary skin hypersensitivity induced by neural provocation and change in conditioned pain modulation after immune provocation; the proxy for vulnerability to fatigue is heart rate variability 24h after immune provocation. Immune responsiveness is represented by IL-6 and TNF-α levels in supernatant after in vitro lipopolysaccharide provocation of whole blood. The investigators hypothesise that levels of IL-6 and TNF-α after in vitro immune provocation will be positively associated with the area of secondary skin hypersensitivity after in vivo neural provocation, and negatively associated with conditioned pain modulation after in vivo immune provocation.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65 years old.

Exclusion Criteria:

* Incompetence to consent and participate, e.g. acute psychosis or high suicide risk.
* Pregnancy,
* Electrical implants (e.g. pace-maker),
* Metal implants in the forearm,
* Tattoos on the forearm,
* Any visible injury or open wounds in the forearm,
* Known history of allergic reactions to vaccines,
* Has received the current season's influenza vaccine,
* Chronic pain (pain on most days for the past 3 months),
* Diabetes Mellitus,
* Peripheral vascular disease,
* Sensory impairment in the forearm, shoulder and lower back,
* Use of medication that could later skin sensitivity (e.g. analgesic medication, immune modulators, topical medical creams),
* Cardiovascular disorders,
* Medication that alters immune function (e.g. NSAIDs, steroids),
* Smoking habit,
* Febrile illness in the preceding 4 weeks.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit healthy adult volunteers (≥18 and ≤ 65 years old) with a range of childhood trauma. All interested volunteers will complete the Childhood Trauma Questionnaire-Short form. The investigators will use the total score on the questionnaire to recruit specifically for a varied range in childhood adversity history and enrol participants into three similarly sized groups: 1) minimal childhood adversity (control) (score 25-36), 2) low-moderate childhood adversity (score 37-67), and 3) severe childhood adversity (score > 67). The investigators will enrol volunteers into each group using a 'first to qualify, book, and attend the testing sessions' approach, with the goal of achieving similar group sizes. Some groups may fill up faster than others.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Childhood Trauma Questionnaire-Short form | Baseline
  The Childhood Trauma Questionnaire-Short form uses 28 statements to probe five domains: emotional abuse, physical abuse, sexual abuse, emotional neglect, and physical neglect. Participants rate the extent to which each of the 28 possible situations was true during their childhood and adolescence, on a 5-point Likert scale ranging from "never true" to "very often true". The total score is computed by summing scores across forward- and reverse-coded items and a separate denial score that is obtained using three of the items. A higher score indicates more childhood adversities (i.e. worse outcome). The investigators will use the total score on the Childhood Trauma Questionnaire-Short to recruit specifically for a varied range in childhood adversity history and enrol participants into three similarly sized groups: 1) minimal childhood adversity (control) (score 25-36), 2) moderate childhood adversity (score 37-67), and 3) severe childhood adversity (score > 67).
Provoked inflammatory response | Baseline
  Mean z-scores of IL-6 and TNF-alpha levels
Secondary hypersensitivity (surface area) | 30 minutes, 45 minutes and 60 minutes after the high-frequency electrical stimulation (neural provocation)
  Surface area of secondary hypersensitivity induced by high-frequency electrical stimulation
Conditioned pain modulation | Baseline and 24 hours after the influenza vaccine (immune provocation).
  Change in pressure pain threshold (test stimulus) after cold water immersion (conditioning stimulus)
Temporal summation | Baseline and 24 hours after the influenza vaccine (immune provocation).
  Mechanical stimuli will be provided from a 256mN von Frey Filament. Participants will provide ratings to mechanical stimuli using the Sensation and Pain Rating Scale. The Sensation and Pain Rating Scale has a 'non-painful' range, on the left of the scale, ranging from -50 - "no sensation" to 0 - "the exact point at which what you feel transitions to pain". The 'painful' range, on the right of the scale, ranges from 0 to +50 - "most intense pain you can imagine". A lower score means less intense sensation/pain (i.e. better outcome) and a higher score means more intense sensation/pain (i.e. worse outcome).

SECONDARY OUTCOMES:
Heart rate variability | Baseline, 40 minutes after the high-frequency electrical stimulation (neural provocation), and 24 hours after the influenza vaccine (immune provocation).
  Using 3-lead ECG and Biopac System
N-back test | Baseline and 24 hours after the influenza vaccine (immune provocation).
  Assessing working memory
6-minute walk test | Baseline and 24 hours after the influenza vaccine (immune provocation).
  Assessing physical exertion and recovery
Secondary hypersensitivity (magnitude) | Baseline, and 35 minutes, 50 minutes and 65 minutes after the high-frequency electrical stimulation (neural provocation).
  Change in ratings on the Sensation and Pain Rating Scale to punctate mechanical stimulation. The Sensation and Pain Rating Scale has a 'non-painful' range, on the left of the scale, ranging from -50 - "no sensation" to 0 - "the exact point at which what you feel transitions to pain". The 'painful' range, on the right of the scale, ranges from 0 to +50 - "most intense pain you can imagine". A lower score means less intense sensation/pain (i.e. better outcome) and a higher score means more intense sensation/pain (i.e. worse outcome).
Static and dynamic light touch, and single electrical stimulation | Baseline, and 35 minutes, 50 minutes and 65 minutes after the high-frequency electrical stimulation (neural provocation)
  Change in ratings on the Sensation and Pain Rating Scale to punctate mechanical stimulation. The Sensation and Pain Rating Scale has a 'non-painful' range, on the left of the scale, ranging from -50 - "no sensation" to 0 - "the exact point at which what you feel transitions to pain". The 'painful' range, on the right of the scale, ranges from 0 to +50 - "most intense pain you can imagine". A lower score means less intense sensation/pain (i.e. better outcome) and a higher score means more intense sensation/pain (i.e. worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Victoria J Madden, PhD, Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
The data management plan complies with the South African Protection of Personal Information Act (POPIA) of 2013. All coded data (from the screening, enrolment and data collection phases) will be stored in a password-protected Google Drive folder, under the governance of the PI. Additionally, the back-up external hard drives will be stored in a secure location.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: In keeping with open science, and following a final assessment to eliminate the possibility of reverse identification of any participant, all coded data will be made publicly available via a public repository (e.g GitHub) at study completion.

REFERENCES:
- [Derived] Bedwell GJ, Mqadi L, Kamerman P, Hutchinson MR, Parker R, Madden VJ. Inflammatory reactivity is unrelated to childhood adversity or provoked modulation of nociception. Pain. 2025 Nov 1;166(11):e590-e605. doi: 10.1097/j.pain.0000000000003658. Epub 2025 May 15. PMID 40372281